CLINICAL TRIAL: NCT04462458
Title: Clinical and Radiological Outcomes of M-ARS ACL
Brief Title: M-ARS ACL Post-marketing Surveillance Study
Status: Recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P07.001.01
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Anterior Cruciate Ligament (ACL) Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Medacta Anatomic Ribbon Surgery (M-ARS ACL) — M-ARS ACL allows to reconstruct the anterior cruciate ligament using the Anatomic Ribbon Technique

SUMMARY:
The goal of this study is to evaluate the performance of Medacta Anatomic Ribbon Surgery (M-ARS) in patients requiring anterior cruciate ligament (ACL) reconstruction.

The main goal is to evaluate the survival rate of M-ARS ACL at 6 months post-operatively. The secondary goals are to assess the survival rate, clinical and functional outcomes, the quality of life, and the rate of complications at 1 month, 1 year and 2 years post-operatively.

DETAILED DESCRIPTION:
This s a prospective, multicenter, non-controlled, observational study to evaluate the outcomes of Medacta Anatomic Ribbon Surgery (M-ARS) in the reconstruction of the anterior cruciate ligament (ACL).

Participants will be informed about the study, both orally and in writing, during a preoperative visit. The investigator will answer any questions that may arise and will collect the informed consent. During the study, enrolled participants will be able to withdraw at any time and for any reason.

The study is conducted according to the following schedule:

* V1 : Inclusion during a preoperative visit
* V2: Surgery
* V3: Follow-up visit at 1 month ± 15 days post-surgery
* V4: Follow-up visit at 6 months ± 30 days post-surgery
* V5: Follow-up visit at 12 months ± 60 days post-surgery
* V6: Follow-up visit at 24 months ± 90 days post-surgery

The following data will be collected:

* Survival rate of implants evaluating the incidence of implants failure, where implant failure is defined as revision, loosening, or any definite change in the position of components (V3-V6).
* Clinical and functional outcomes, measured with the International Knee Documentation Committee (IKDC) score (V1, V3-V6)
* Quality of Life, measured with the EQ-5D score (V1, V3-V6)
* Occurrence of intraoperative and postoperative complications (V2-V6)

Depending on standard practice, imaging assessment of implants and bone tunnels may be performed.

A web-based data collection tool will be used as Electronic Data Capture (EDC). All the information required by the protocol will be collected in electronic case report forms (eCRF).

The statistical analysis will be performed according to a pre-established statistical analysis plan. Missing values will not be replaced by estimated values but will be considered as missing in the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients with ACL rupture requiring ACL reconstruction

Exclusion Criteria:

* Patients with malignant diseases (at the time of surgery)
* Patients with proven or suspected infections (at the time of surgery)
* Patients with functional deficits of the affected extremity (at the time of surgery)
* Patients with known incompatibility or allergy to products materials (at the time of surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring ACL reconstruction and who are suitable to receive M-ARS ACL will be proposed to take part to the current post-marketing surveillance study during their pre-operative visit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 6 months
  Kaplan Meier method

SECONDARY OUTCOMES:
Survival rate | 1, 12, 24 months
  Kaplan Meier method
Functional outcome | 1, 6, 12, 24 months
  International Knee Documentation Committee (IKDC) score
Quality of Life outcome | 1, 6, 12, 24 months
  EQ-5D score
Radiological outcome (optional) | 1, 6, 12, 24 months
  Evaluation of ligament osteointegration, femoral/tibial tunnel widening, presence of fluid in the femoral/tibial tunnel
Complication rate | intraoperative, 1, 6, 12, 24 months
  Occurrence of intraoperative and postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Mirco Herbort, Prof. Dr. med., Principal Investigator — OCM Klinik GmbH
Locations (3):
- Austria (2):
  - Praxis Gelenkpunkt - Sport- und Gelenkchirurgie, Innsbruck
  - Pyhrn-Eisenwurzen Klinikum Kirchdorf, Kirchdorf an der Krems
- OCM Klinik GmbH, München, Germany